CLINICAL TRIAL: NCT03895463
Title: Prospective Noninterventional Study to Assess the Use of Lanreotide Autogel® 120 mg in Patients With Locally Advanced or Metastatic Gastroenteropancreatic Tumours (GEP-NETs) in Routine Clinical Practice
Brief Title: Study to Assess the Use of Lanreotide Autogel® 120 mg in Patients With Locally Advanced or Metastatic Gastroenteropancreatic Neuroendocrine Tumours (GEP-NETs) in Routine Clinical Practice
Acronym: NETways
Status: Withdrawn | Type: Observational
Why Stopped: Reassessment of study feasibility
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-PL-52030-380
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this study is to assess the Progression-Free Survival (PFS) at 12 months of Lanreotide Autogel 120 mg use when administered as part of routine GEP-NET treatment and to follow patient treatment pathways, identify prognostic factors of PFS, evaluate patient's QoL, and patient's and clinician's satisfaction with treatment in routine long-term care setting. The study will provide real-world evidence on the use of Lanreotide Autogel 120 mg and will provide information on topics such as optimization of product usage and identification of best practices and will provide evidence on product effectiveness in a realistic setting.

ELIGIBILITY:
Inclusion Criteria:

* Functioning or non-functioning histopathologically confirmed, locally advanced or metastatic (grade 1 or grade 2 according to the World Health Organisation (WHO) 2017 classification and European Neuroendocrine Tumour Society (ENETS) grading system) GEP-NET G1,G2 (Ki67≤10%, based on recent Ki67).
* Measurable disease, as defined by RECIST 1.0, on a CT scan/MRI obtained up to 6 weeks prior to initiation of treatment with Lanreotide Autogel 120 mg.
* Subject eligible for treatment with Lanreotide Autogel 120 mg or subject currently being treated with Lanreotide Autogel 120 mg administered every 28 days for a period no longer than 5 months prior to inclusion
* Treatment with Lanreotide Autogel 120 mg alone, according to local Summary of Product Characteristics (SmPC).

Exclusion Criteria:

* Lanreotide Autogel treatment for more than 5 months prior to inclusion into the study
* Concomitant anti-proliferative medication/therapies for GEP NET at initiation of Lanreotide Autogel treatment (e.g. Peptide Receptor Radionuclide Therapy (PRRT), cytotoxic chemotherapy, targeted therapy everolimus, sunitinib, interferon, loperamide).
* Has been treated with PRRT, chemotherapy, everolimus, sunitinib or interferon within 3 months prior to initiation of Lanreotide Autogel treatment
* Parallel participation in an interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with GEP-NETs eligible for treatment with Lanreotide Autogel 120 mg or currently being treated with Lanreotide Autogel 120 mg every 28 days for a period of up to 5 months. Subjects will receive treatment as prescribed by the physician and in accordance with the current Summary of Product Characteristics (SmPC).
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2023-03-26 (Estimated); Study Completion 2023-03-26 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 12 months
  To estimate the rate according to investigator assessment (radiological progression; based on Response Evaluation Criteria In Solid Tumours version 1.0 [RECIST 1.0])

SECONDARY OUTCOMES:
Median PFS | 24 months
Tumour origin | 24 months
Tumour grade | 24 months
Quality of Life (QoL) | 24 months
  To describe the change in Quality of Life (QoL) as assessed by European Organisation for Research and Treatment of Cancer (EORTC) QoL questionnaire for gastrointestinal neuroendocrine tumours (QLQ-GINET21 questionnaires). Where the patient assess experienced symptoms or problems using the scale from 1 to 4. Where 1 represents "not at all" and 4 "very much".
Disease Control Rate | 24 months
  To estimate the Disease Control Rate (DCR), as assessed by investigator (proportion of subjects with a best overall response of Partial Response [PR], Complete Response [CR] or Stable Disease [SD]).
Chromogranin A (CgA) level | 24 months
Patients' satisfaction | 24 months
  To evaluate patients' satisfaction using abbreviated 9-item Treatment Satisfaction Questionnaire for Medication (TSQM-9). It assesses key dimensions of treatment satisfaction: Effectiveness, Convenience and Global Satisfaction. The effectiveness scored as: 1 (extremely dissatisfied) to 7 (extremely satisfied). For the convenience scored as 1 (extremely difficult) to 7 (extremely easy).
Urine 5-hydroxyindoleaceticacid (5-HIAA) levels | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (11):
- Poland (11):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Oddział w Gliwicach, Gliwice
  - Uniwersyteckie Centrum Kliniczne im. Prof. K. Gibińskiego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Świętokrzyskie Centrum Onkologii, Kielce
  - Szpital Uniwersytecki w Krakowie, Krakow
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - Szpital Kliniczny im. Heliodora Święcickiego Uniwersytetu Medycznego w Poznaniu, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 Pomorskiego Uniwersytetu Medycznego im. prof. Tadeusza Sokołowskiego, Szczecin
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie, Warsaw
  - Uniwersyteckie Centrum Kliniczne Warszawskiego Uniwersytetu Medycznego, Centralny Szpital Kliniczny, Warsaw
  - Dolnośląskie Centrum Onkologii we Wrocławiu, Wroclaw